CLINICAL TRIAL: NCT06109896
Title: ONCO_STORIES. Stress, Trauma, Origins, Psychological Responses, Interpersonal Relationships and Experiences in the Clinical History of Cancer Patients
Brief Title: Clinical Stories and Psychological Experiences of Cancer Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 5913
Record Dates: First submitted 2023-10-26; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Tumor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Self Report Questionaires — Collection and analysis of information from patient self-report assessments and integration with clinical information from assessments performed routinely during cancer treatment.

SUMMARY:
The purpose of the study is to collect and analyze information from the multidimensional assessment of cancer patients (medical, psychological, psychometric, biological, etc.) treated at the Fondazione Policlinico Universitario Agostino Gemelli IRCCS. The collection of information will allow to investigate the possible presence of correlations between psychological aspects and clinical medical conditions of the person during the course/treatment of cancer.

In the course of the study, the possible presence of previous stressful and/or traumatic events, and the presence of psychological, post-traumatic and/or dissociative symptoms during treatment will be explored. Any correlations between medical conditions and psychological, emotional and behavioral characteristics will also be explored. Finally, it will be possible to investigate the effectiveness of psychological interventions that are carried out according to clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between 18 and 99 years old;
* Individuals with a diagnosis of current oncologic disease and in active oncologic treatment at the hospital where the study is conducted;
* Individuals with a history of oncologic disease who have completed oncologic treatment or in follow-up at the hospital where the study is conducted;

Exclusion Criteria:

* Non-signing of informed consent;
* Non-signing of consent/assent by patient/legal guardian;
* Patients with cognitive impairment or legal disqualification;
* Clinical/medical or psychological condition that does not allow completion of self-report questionnaires;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who have been diagnosed with cancer. Patients who access the services of: Gynecology Oncology Unit, Internal Medicine and Gastroenterology Unit, Digestive Surgery Unit, Radiotherapy Oncology Unit, Senology Surgery Unit, Medical Oncology Unit, Hematology Unit, Medicine Unit will be considered.
  Neurosurgery and at the same time as psychological consultation with the operators belonging to the Clinical Psychology Unit of Fondazione Policlinico Universitario A. Gemelli IRCSS.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-10-31 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Collect and analyze information from the multidimensional assessment of cancer patients | 1 hour
  Descriptive and statistical analysis of data collected on the clinical and psychological conditions of the cancer patient through routine assessments and self-report questionnaires.